CLINICAL TRIAL: NCT01928420
Title: A Single Site, Randomized, Double-blind, Placebo Controlled Trial of NIC5-15 in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT01928420; R21AT003302-01A1 (NIH); MHBB-009-06S (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2012-08-17; First posted 2013-08-26 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer Disease; Alzheimer Type Senile Dementia; Alzheimer's Disease; clinical trial; dementia; diabetes; dietary supplements; Senile Dementia, Alzheimer; Therapeutics; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Delirium, Dementia, Amnestic, Cognitive; Disorders; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Diabetes Mellitus; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Delirium; Disease; Mental Disorders | interventions — pinitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIC5-15 (Experimental): Subjects with Alzheimer's Disease Intervention: Drug: NIC5-15
  Interventions: Drug: Drug: NIC5-15
- Placebo (Placebo Comparator): Subjects with Alzheimer's Disease Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: NIC5-15 — A natural product, found in many foods and plants with mild insulin sensitizing effects
  Other Names: Pinitol
  Arms: NIC5-15
Drug: Placebo — Subjects with Alzheimer's Disease placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NIC5-15 in the treatment of Alzheimer's Disease.

DETAILED DESCRIPTION:
Recent epidemiologic evidence, has suggested that diabetes mellitus significantly increases risk for the development of Alzheimer's disease, independent of vascular risk factors. Moreover, even patients who are simply insulin resistant, without frank diabetes, have been shown to share this elevated risk for the development of AD. As insulin's role as a neuromodulator in the brain has been revealed, several potential mechanisms for the interaction of diabetes or insulin resistance with AD have been suggested such as decreased cortical glucose utilization particularly in the hippocampus and entorhinal cortex; increased oxidative stress through the formation of advanced glycation end products; increased Tau phosphorylation and neurofibrillary tangle formation; and increased beta-amyloid aggregation through inhibition of insulin-degrading enzyme. The future treatment of AD might involve pharmacologic and dietary manipulations of insulin and glucose regulation

NIC5-15 is a single, small, naturally occurring molecule. Animal studies and some human trials have shown NIC5-15 to be safe and a potent insulin sensitizer at doses equivalent to 800-2000mg per day. In preclinical studies at doses higher than those previously studied in clinical trials, we found that NIC5-15 interferes with the accumulation of beta amyloid, an important step in the development of Alzheimer's pathology. These data suggest that NIC5-15 may be a reasonable therapeutic agent for the treatment of Alzheimer Disease for two reasons:

It is a -secretase inhibitor that is Notch-sparing. It is potentially an insulin-sensitizer.

However critical safety and human efficacy studies must be conducted. This application proposes to conduct these early critical human studies. The goal of the studies contained in this proposal is to establish safety and efficacy of NIC5-15 for the treatment of AD. The specific objectives of this study are to:

Specific Objective #1) Conduct a multiple dose safety study of NIC5-15 to establish safety in the doses that appear to block amyloid accumulation. These studies will characterize the safety profile, pharmacokinetics, and tolerability

This objective was met with completion of the initial study ID#NCT00470418.

The current study continues investigations of NIC5-15 in Alzheimer's disease with the following objective:

Specific Objective #2) Conduct a double blind placebo controlled pilot efficacy study of NIC5-15 in patients with AD. The goals of this study are to:

A) Demonstrate feasibility for a multi-site trial that will be used to guide the design of a future larger effort. Demonstration of feasibility will include examination of accrual rate, overall recruitment, adherence to protocol, compliance with medication and willingness to complete a randomized trial, and lack of short term toxicity.

B) Collect preliminary evidence of efficacy in terms of cognitive and global measures as well as secondary efficacy outcomes of activities of daily living, behavioral disturbances and AD biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* NINCDS/ADRDA criteria for probable AD
* MMSE between 12-27
* Treatment with a cholinesterase inhibitor or an NMDA (N-methyl-D-asparate) antagonist with stable dose for at least 12 weeks
* Home monitoring available for supervision of medications
* Caregiver available to accompany patient to all visits and willing to participate in study as informant
* Fluent in English or Spanish
* Medical stability for this study as confirmed by review of records, internist's physical exam, neurological exam, and laboratory tests
* Stable doses of non-excluded medication
* No evidence of hepatic insufficiency
* Able to swallow oral medications
* Ability to participate in the informed consent process

Exclusion Criteria:

* History of Diabetes Mellitus (OGTT criteria) requiring treatment with an excluded antidiabetic medication (see below) or history of hypoglycemia
* Active hepatic or renal disease
* Cardiac disease including history of congestive heart failure or current treatment for CHF; history of recent myocardial infarction
* Use of another investigational drug within the past two months
* History of clinically significant stroke
* History of seizure or head trauma with disturbance of consciousness within the past two years
* Major mental illness including psychotic disorders, bipolar disorder, or major depressive episode within the past two years Medication Exclusion
* Current use of oral hypoglycemic agents including sulfonylureas and meglintinides
* Current or past treatment with insulin for longer than two weeks
* Current use of drugs with significant anticholinergic or antihistaminic properties

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)Score | Over 6 months, measured at visits 2 (week 2), 6 (week 12), 8 (week 24)
  A psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Cooperative Study Clinician's Global Impression of Change (ADCS-CCGIC) Score | Over 6 months, measured at visits 2 (week 2), 6 (week 12), 8 (week 24)
  A systematic method for assessing clinically significant change in a clinical trial as viewed by an independent skilled and experienced clinician . The ADCS-CGIC focuses on clinician's observations of change in the subject's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the subject and an interview of an informant. Unlike a targeted symptom scale, it takes into account a subject's overall function in the cognitive, behavioral, and functional activity domains.
Change in Mini-Mental State Examination (MMSE) Score | Over 6 months, measured at visits 2 (week 2), 6 (week 12), 8 (week 24)
  A frequently used screening instrument for Alzheimer's disease drug studies. It evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) Score | Over 6 months, measured at visits 2 (week 2), 6 (week 12), 8 (week 24)
  ADCS-ADL assesses functional performance in subjects with Alzheimer's disease. In a structured interview format, informants are queried as to whether subjects attempted each item in the inventory during the prior 4 weeks and their level of performance. The ADCS-ADL scale discriminates well between normal controls and mild AD patients. It has good test-retest reliability. The ADCS-ADL includes some items from traditional basic ADL scales (e.g., grooming, dressing, walking, bathing, feeding, toileting) as well as items from instrumental activities of daily living scales (e.g., shopping, preparing meals, using household appliances, keeping appointments, reading).
Change in Neuropsychiatric Inventory (NPI) Score | Over 6 months, measured at visits 2 (week 2), 6 (week 12), 8 (week 24)
  The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology and behavior in AD based on interview with the informant.
Changes in AD Biomarkers | Blood collected at visits 2 (week 2), 6 (week 12), 8 (week 24)
  Plasma beta-amyloid proteins will be collected from blood samples obtained at visit 2 (week 2), visit 6 (week 12), and visit 8 (week 24).
APO-E genotyping | Collected at visit 2 (week 2)
  APOe e4 is an important genetic risk factor for AD. In this trial, as in many studies of AD and memory and cognition in aging, the APOe e4 allele will be analyzed as a predictor of clinical change over time.

OTHER OUTCOMES:
Symptoms Checklist and Adverse Event Assessment | 6 Months, conducted at visits 3 (week 2), 4 (week 4), 5 (week 8), 6 (week 12), 7 (week 18), 8 (week 24)
  Adverse events and symptoms checklist are used to monitor signs or symptoms that may or may not be related to study medication, abnormalities detected during physical examination, or clinical significant laboratory abnormalities.
Safety Laboratory Assessments | 6 Months, conducted at visits 1 (week 1), 3 (week 2), 4 (week 4), 5 (week 8), 6 (week 12), 7 (week 18), 8 (week 24)
  Blood tests: hematology, serum chemistries, folate, B12, RPR, thyroid function (TSH or free thyroxine index), Urinalysis, Metabolic panel: HgbA1c, triglyceride profile serum albumin
Neurological examination | 6 Months, conducted at visits 1 (week 1), 6 (week 12), 8 (week 24)
  Neurological examination measuring any possible sensory impairments and/or neurological abnormalities to determine if findings are consistent with eligibility for safety. This must be signed by a clinician.
Physical examination | 6 Months, conducted at visits 1 (week 1), 3 (week 2), 5 (week 8), 6 (week 12), 7 (week 18), 8 (week 24)
  Standard physical examination of vital signs, weight and height (to calculate BMI), seated blood pressure, EKG, seated pulse rate, respiration rate, and temperature, to determine if findings are consistent with eligibility for safety, which must be signed by a clinician.
Pharmacokinetic analysis | 6 Months, conducted at visits 2 (week 2), 8 (week 24)
  A single assay of NIC5-15 concentration in blood samples obtained at visit 2 (week 2) and visit 8 (week 24).

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Grossman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J Peters Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided